CLINICAL TRIAL: NCT03349086
Title: Effects of Vocal Exercise Following Botox Injection on Voice Handicap and Communicative Participation for Adductor Spasmodic Dysphonia
Brief Title: Effects of Vocal Exercises for Spasmodic Dysphonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-1746
Record Dates: First submitted 2017-08-31; First posted 2017-11-21 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Adductor Spasmodic Dysphonia
Keywords: Botox Injection; Spasmodic; Dysphonia; Voice Therapy; Speech Therapy; Voice Rest
MeSH Terms: conditions — Dysphonia; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Participants will undergo one of two study conditions immediately following a standard of care Botox injections. One condition is a 45 minute voice rest condition and the other condition is a 45 minute voice exercise condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice Exercise (Active Comparator): Randomized participants in this group will undergo 45 minutes of voice exercise, including sustained pitches and pitch glides on a variety of different vocal facilitators.
  Interventions: Behavioral: Voice Exercise
- Voice Rest (No Intervention): Randomized participants in this group will undergo 45 minutes of voice rest.

INTERVENTIONS:
Behavioral: Voice Exercise — Voice exercise will consist of sustained pitches and pitch glides on a variety of different vocal facilitators.
  Arms: Voice Exercise

SUMMARY:
The purpose of this study is to assess the effect of voice exercise and voice rest on subject's perception of vocal handicap and communicative participation following Botox injections for adductor spasmodic dysphonia.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD) is a neurological disorder characterized by involuntary spasms of the vocal folds resulting in a strained and strangled voice quality. This disorder is quite disabling to patients who suffer from it, particularly affecting patients' quality of life. Botulinum toxin (Botox) has been found to be the most effective treatment for SD. The Botox is injected into the affected muscle resulting in temporary weakening of the muscle. The patients return for injections on average every 3 - 6 months.

There is a suggestion in the literature that increased diffusion of the Botox injectate could improve the effects of the injection. Furthermore, there is literature supporting the use of exercise to increase the diffusion of the Botox. Previous research examined the use of voluntary muscle activity vs. rest immediately following Botox injection for writer's cramp. It was found that the active condition resulted in greater reduction of muscle strength in the injected muscle. Another small study of 9 patients implemented intense exercise comprised of loud reading for one hour and a rest condition of total voice rest for 24 hours. They found that the exercise condition resulted in improved scores on the voice related-quality of life (V-RQOL) measure and concluded that improvement in results of Botox injections may be achieved more consistently with the implementation of exercise following the injection. The exercise used in this study was intense and may be contrary to the overall benefit as the subjects may experience phonotrauma. Timing of the exercise post-injection may also be a factor. Previous literature review revealed combined modality treatment of Botox injection only, Botox with therapy and Botox with sham treatment. They found no significant differences in acoustic stability, V-RQOL, or duration of injection benefit. However, the exercise was initiated 3 weeks post-injection and completed once per week for 5 weeks. Investigators aim to identify what might improve or extend the duration of botox injections for adductor Spasmodic dysphonia.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 21-70 age
3. Diagnosed with pure adductor spasmodic dysphonia
4. Completed 2 consecutive standard of care Botox injection into the thyroarytenoid (TA) and/or thyroarytenoid/lateral cricoarytenoid (TA/LCA) junction with the same dosage

Exclusion Criteria:

1. Receiving Botox to other laryngeal or supraglottic musculature
2. Other neuro-laryngological conditions
3. Those with an average of less than two injections per year

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
A quantifiable difference between the effects of voice exercise vs. voice rest post Adductor Spasmodic Dysphonia botox treatment through analysis of the Voice Handicap Index Questionnaire. | Assessing the change of the post VHI questionnaire between groups. Data will be reported at study completion, an average of 1 year.
  Pre randomized condition and post 6 week and 12 week, participants will be asked to complete the Voice Handicap Index (VHI).
  The VHI Questionnaire (Voice Handicap Index) is a 30-item questionnaire divided into 3 subsections (Functional, Physical, Emotional) and a Total which measures the effect of voice problems on quality of life. Individuals mark each item on this 30-item questionnaire on a scale from 0-4 (0 being never and 4 being always). Points for each subscale are tallied and a total composite score is also given. A total score of 0-11 is considered Normal, 12-28 is considered Mild Minimal handicap, 29-56 is considered Moderate Handicap, and 57-120 is considered severe handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Brienne Ruel, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No